CLINICAL TRIAL: NCT06907316
Title: Cefixime Versus Benzathine Penicillin G in Treatment of Early Syphilis - a Randomized, Multicentre, Non-inferiority, Open Label Trial
Brief Title: Cefixime Versus Benzathine Penicillin G in Treatment of Early Syphilis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: For financial and personnel reasons, patient recruitment was carried out in only one of the planned centers.
Sponsor: Bulovka Hospital (Other)
Collaborators: Všeobecná fakultní nemocnice Praha (Unknown); Národní referenční laboratoř pro syfilis, Státní zdravotní ústav (Unknown); Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Filip Rob MD, PhD, Chair of Department, Bulovka Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.6.2021/10071/EK-Z
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Syphilis
Keywords: syphilis; treatment; cefixime
MeSH Terms: conditions — Syphilis | interventions — Cefixime

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cefixime (Experimental): cefixime 400 mg taken orally two times a day for 14 consecutive days
  Interventions: Drug: Cefixime 400mg
- benzathine penicillin G (Active Comparator): benzathine penicillin G 2.4 MIU single dose intramuscularly
  Interventions: Drug: Benzathine penicillin 2.4 million units

INTERVENTIONS:
Drug: Cefixime 400mg — cefixime 400 mg taken orally two times a day for 14 consecutive days
  Arms: Cefixime
Drug: Benzathine penicillin 2.4 million units — single dose of benzathine penicillin G 2.4 MIU intramuscularly
  Arms: benzathine penicillin G

SUMMARY:
This study evaluates the efficacy (non-inferiority) and safety of a new antibiotic treatment (cefixime), which has been previously used for single dose therapy of gonorrhoea in many years , in the treatment of early syphilis. Participants will be randomized to one of two study arms and will receive either expirimental regimen (cefixime) or the current standard antibiotic regimen (benzathine penicillin G). New treatment alternatives for syphilis could ensure that people are appropriately treated during periods or in settings of benzathine penicillin G stock out, penicillin allergy, or other intolerance to penicillin injection. This study may also identify an oral regimen for settings in which injections are not feasible.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Non-pregnant, non breastfeeding
3. Able to provide informed consent
4. Clinically or laboratory-confirmed primary, secondary or early latent syphilis with a positive rapid treponemal test and an RPR/VDRL titer equal to or greater than 1:8
5. Non-cephalosporin allergic
6. Non-penicillin allergic
7. Agree to be occasionally called by study staff to be reminded to take study drug
8. Willing to attend follow-up visits

Exclusion Criteria:

1. Under 18 years of age
2. Pregnancy, breastfeeding
3. Prior history of syphilis in last two years
4. Allergy or contraindication to penicillin or cephalosporins (including allergy to cefixime)
5. Systemic antibiotic therapy in last two weeks
6. Previous enrollment in the study
7. Presenting a situation or condition that would not allow reliable study follow up (For example: frequent travel, alcohol abuse or substance misuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Serological cure | from baseline (treatment) to 3 months after treatment
  a 4-fold or more (≥2 dilution steps) decrease in rapid plasma reagin (RPR) or veneral disease reach laboratory test (VDRL) titer

SECONDARY OUTCOMES:
Secondary serological cure | from baseline (treatment) to 6 and 12 months after treatment
  a 4-fold or more (≥2 dilution steps) decrease in rapid plasma reagin (RPR) or veneral disease reach laboratory test (VDRL) titer
Treatment safety | from baseline till the end of follow-up (12 months from baseline)
  Occurrence of treatment-related severe adverse events in treatment groups

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Národní referenční laboratoř pro syfilis, Státní zdravotní ústav, Prague
  - Fakultní nemocnice Bulovka, Prague

IPD SHARING:
Plan to Share IPD: No